CLINICAL TRIAL: NCT02970201
Title: Improving Adherence in Renal Dialysis Patients; a Randomized Crossover Trial for an Electronic Intervention
Brief Title: Improving Adherence in Renal Dialysis Patients Through Electronic Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Will R Ross, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 201412068
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Endstage Renal Disease
Keywords: eHealth; mHealth; Hemodialysis; Adherence; Electronic intervention; ESRD; Nephrology
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period I EpxDialysis (SMS Messaging) (Other): SMS Messaging arm receives the intervention (EpxDialysis) first, then resumes standard of care at crossover (8 weeks).
  Interventions: Other: EpxDialysis
- Period II EpxDialysis (Control) (Other): Control arm receives standard of care first, then receives the intervention (EpxDialysis) at crossover.
  Interventions: Other: EpxDialysis

INTERVENTIONS:
Other: EpxDialysis — The EpxDialysis intervention consists of automated SMS text or voice messages delivered to the patient's preferred phone number three times per week. These messages provide details about the subject's upcoming hemodialysis session, anticipatory guidance regarding clinically-concerning symptoms, as well as the option for direct call routing to the dialysis center for rescheduling sessions.

SUMMARY:
Dialysis treatment non-adherence is a prevalent problem among the end-stage renal population receiving chronic hemodialysis. The complications associated with missed or shortened dialysis sessions are serious and frequently require emergent medical care or hospitalization. Previous studies have shown that electronic messages have significantly improved attendance rates in a primary care setting, but these messages have not been validated in the chronic dialysis population.

An electronic intervention has been developed by Epharmix, a WUSTL IDEA Labs (ideas.wustl.edu) team, which has the capacity to use automated SMS text messages and/or phone calls to notify patients prior to each upcoming appointment, as well as alert a designated patient advocate. Patients receiving the messages are provided with key contact information for a dialysis rescheduling phone line, transportation resources, social work services, etc. They may also receive instructions on what to do if they are experiencing physical symptoms and need educational facts about dialysis. In particular, the intervention is designed to demonstrate to patients that the center cares and is concerned for their health and wellbeing. This intervention may potentially improve patient adherence to their scheduled sessions, increase patient satisfaction with their treatment, and prevent medical complications associated with missed dialysis appointments.

This study aims to determine whether an electronic intervention, which sends SMS text messages or phone calls of key dialysis treatment information, is able to improve dialysis treatment session attendance among dialysis patients with a history of poor attendance. We secondarily aim to identify the factors that may be barriers to dialysis treatment session attendance and the emergency department or hospital utilization associated with missed dialysis treatments.

Patients will be prospectively identified, recruited, and randomized into two groups. Group A will receive the electronic intervention prior to their appointments; Group B will not receive any electronic intervention. After 8 weeks, crossover will occur for both groups and the study will continue for an additional 8 weeks. Participants' clinic records will be reviewed to determine the numbers of missed and attended appointments, as well as records of ED visits and hospital admissions. Subjects will be asked to complete a post-study satisfaction questionnaire.

DETAILED DESCRIPTION:
Dialysis treatment non-adherence is a prevalent problem among the end-stage renal population receiving chronic hemodialysis. The complications associated with missed or shortened dialysis sessions are serious and frequently require emergent medical care or hospitalization. Previous studies have shown that electronic messages have significantly improved attendance rates in a primary care setting, but have not been validated in the chronic dialysis population.

An electronic intervention has been developed by Epharmix, a WUSTL IDEA Labs (ideas.wustl.edu) team, which has the capacity to use SMS text messaging to phone call recordings to notify patients prior to each of their upcoming appointment times, with the option of also alerting a designated patient advocate. Patients receiving the messages are provided with key contact information for a dialysis rescheduling phone line, transportation resources, social work services, etc. This intervention may potentially improve patient adherence with scheduled sessions, increase patient satisfaction with their treatment and prevent medical complications associated with missing dialysis.

This study aims to determine whether an electronic intervention, which sends SMS text messages or phone calls of key dialysis treatment information, is able to improve dialysis session attendance among patients with a history of poor attendance. Our secondary aim is to identify factors that may be barriers to dialysis appointment attendance and are associated with emergency department (ED) or hospital utilization.

Procedures: Dialysis patients of the Chromalloy American Kidney Center (CAKC) at Barnes Jewish Hospital (BJH) and the Washington University Dialysis Center (WUDC) will be included in this study. Two cohorts will be prospectively identified, one group consisting of individuals with a history of occasional non-attendance to treatment sessions, defined as 2-3 missed sessions out of 24 consecutive sessions in the past 8 weeks; the other group consisting of individuals who are frequently non-adherent (4-6 missed sessions in the past 24 consecutive sessions). Patients from each cohort will be recruited and then randomized to either the experimental or the control group. Group A will receive the electronic intervention featuring automated SMS text message and/or phone call prior to their appointments; Group B will not receive any electronic intervention. After 8 weeks, crossover will occur for both groups and the study will continue for an additional 8 weeks.

At time of enrollment, all subjects will be asked to complete a questionnaire to determine the demographic characteristics of the study population of interest and identify possible socio-economic factors contributing to non-adherence to the prescribed 3 times weekly dialysis schedule. The participants' clinic records will be reviewed to determine the numbers of missed and attended appointments, as well as records of ED visits and hospital admissions through BJH. Subjects will be asked to complete a post-questionnaire to rate their satisfaction with their current schedule of dialysis and their satisfaction with the electronic intervention.

ELIGIBILITY:
Inclusion Criteria:

* All potential subjects are between 18 and 75 years of age, and have been receiving hemodialysis treatments, scheduled for 3 sessions/week, for at least 8 weeks at the Chromalloy American Kidney Center or Washington University Dialysis Center.
* The individuals will be prospectively identified as whether they have a history of occasional non-attendance to dialysis treatments, defined as 2-3 missed appointments in the preceding 8 week period or 24 scheduled sessions. These subjects will be enrolled as part of one cohort. Individuals who have frequent non-attendance, defined as 4-6 missed appointments in the preceding 8 week period or 24 scheduled sessions, will be enrolled as a second cohort.
* Subjects must be able to provide a phone number at which they can either receive SMS text messages and/or phone calls. The cost of messages will be paid for by the sender. Subjects must be able and willing to provide consent and authorize access of their medical record and dialysis clinic record for study use.

Exclusion Criteria:

* Persons not receiving ongoing hemodialysis treatments or new patients with less than 8 weeks of treatments at the dialysis center.
* Persons not intended to receive 3 dialysis treatments/week for the next 8 weeks.
* Pregnant individuals.
* Persons unable to be contacted by phone call or SMS text message, or unwilling to provide their contact number.
* Persons unwilling to consent and follow the assigned regimen and complete the required follow up.
* Persons with severe neurological or cognitive disorders, limiting their ability to provide consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Dialysis appointment attendance | 16 weeks
  The primary objective of this prospective randomized control study is to assess the effects of an electronic intervention, which sends automated SMS text messages or pre-recorded phone messages, on attendance rate to dialysis sessions among non-adherent dialysis patients.

SECONDARY OUTCOMES:
Hospitalization | 16 weeks
  Compare the number of emergency department visits and hospitalizations between groups during intervention and control phases

CONTACTS AND LOCATIONS:
Overall Officials: Will R Ross, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine - Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Renal Data System Annual Data Report. Chapter 1: Incidence, prevalence, patient characteristics and modality. National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD https://www.usrds.org/2015/view/v2_01.aspx (2015)
- [Background] Lamping, D. L. & Campbell, K. A. Hemodialysis Compliance: Assessment, Prediction, and Intervention: Part I. Seminars in dialysis 3, 52-56 (1990).
- [Background] Sherman RA, Cody RP, Matera JJ, Rogers ME, Solanchick JC. Deficiencies in delivered hemodialysis therapy due to missed and shortened treatments. Am J Kidney Dis. 1994 Dec;24(6):921-3. doi: 10.1016/s0272-6386(12)81061-4. PMID 7985669
- [Background] Lamping, D. L. & Campbell, K. A. Hemodialysis Compliance: Assessment, Prediction, and Intervention: Part II. Seminars in dialysis 3, (1990).
- [Background] Cummings KM, Becker MH, Kirscht JP, Levin NW. Intervention strategies to improve compliance with medical regimens by ambulatory hemodialysis patients. J Behav Med. 1981 Mar;4(1):111-27. doi: 10.1007/BF00844851. PMID 7288877
- [Background] Parikh A, Gupta K, Wilson AC, Fields K, Cosgrove NM, Kostis JB. The effectiveness of outpatient appointment reminder systems in reducing no-show rates. Am J Med. 2010 Jun;123(6):542-8. doi: 10.1016/j.amjmed.2009.11.022. PMID 20569761
- [Background] Junod Perron N, Dao MD, Righini NC, Humair JP, Broers B, Narring F, Haller DM, Gaspoz JM. Text-messaging versus telephone reminders to reduce missed appointments in an academic primary care clinic: a randomized controlled trial. BMC Health Serv Res. 2013 Apr 4;13:125. doi: 10.1186/1472-6963-13-125. PMID 23557331
- [Background] Bame SI, Petersen N, Wray NP. Variation in hemodialysis patient compliance according to demographic characteristics. Soc Sci Med. 1993 Oct;37(8):1035-43. doi: 10.1016/0277-9536(93)90438-a. PMID 8235736